CLINICAL TRIAL: NCT03696446
Title: E-health Intervention for Cardiac Rehabilitation: Pilot Implementation and Feasibility
Brief Title: E-health Intervention for Cardiac Rehabilitation
Acronym: VCRP-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VCRP-RCT
Record Dates: First submitted 2018-04-17; First posted 2018-10-04 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Coronary Heart Disease; Valve Disease, Heart
Keywords: Cardiac Rehabilitation; Patient Activation
MeSH Terms: conditions — Coronary Disease; Heart Valve Diseases; Patient Participation

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The facilitators will not know that the participants are part of the study. Participants will know which group they are allocated to as they are aware of both groups (described in the consent form).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Cardiac Rehabilitation Program (Experimental): This group will receive access to the NWC (NexJ Connected Wellness TM (NCW) and will be provided with a fitness tracker (Garmin Vivofit 3) to monitor their exercise, sedentary behaviours, and sleep patterns. The NWC platform includes components for education (health library, workbooks etc), collaboration (personal care plan, appointment scheduler, secure messaging system etc), and motivation (motivational messages on their homepage etc). With the Health Coach, participants will engage in: reviews of their risk factor profile and health priorities; goal setting and action planning; problem solving and skill building; and discussions of relapse prevention. Participants will receive a total of seven hours of health coaching delivered across nine sessions over a 26-week period
  Interventions: Behavioral: Virtual Cardiac Rehabilitation Program
- Case Managed Home Program (Other): The Case Managed Home Program (CMHP) is delivered primarily via telephone. Following their CR intake, patients are linked with their CMHP Health Coach and attends their visit (in person or over the phone) which includes a comprehensive review of their health history, current symptoms, medications, activity, and individual concerns. Following this visit, participants will receive a total of 10 individualized telephone calls over a 26 week period. The program action plan is individually formulated based on the participant's goals and learning needs. Participants are provided with educational kits (exercise, nutrition, stress management or prevention) that are based on the principle of single point learning and incorporate behavioural change techniques.
  Interventions: Behavioral: Case Managed Home Program

INTERVENTIONS:
Behavioral: Virtual Cardiac Rehabilitation Program — This group will receive their Rehab program primarily online through a secure web-based platform with a trained facilitator.
  Other Names: Web-based CR
  Arms: Virtual Cardiac Rehabilitation Program
Behavioral: Case Managed Home Program — This group will receive their Rehab program over the phone with a trained facilitator
  Other Names: Phone based CR
  Arms: Case Managed Home Program

SUMMARY:
Cardiac rehabilitation (CR) is designed to increase healthy behaviours (e.g. physical activity, healthy eating, smoking abstinence) and reduce risk factors (e.g. high blood pressure & cholesterol) in order to improve quality of life and health among people with heart disease. Unfortunately, few patients attend CR, often reporting several barriers to access including travel distance, parking fees and lack of time. Advances in technology have the potential to improve accessibility and delivery of CR programs, and improve patient empowerment. The University of Ottawa Heart Institute has developed an e-health program called the Virtual Cardiac Rehabilitation Program (VCRP); an online cardiovascular health management system (website & Smartphone app) that provides strategies for the control and management of risk factors. The goals of VCRP are to: empower and educate patients; foster better communication between patients and their health care team; stimulate shared decision making; and, facilitate care coordination leading to better health outcomes. The VCRP provides patients with: real-time access to their health information, as well as tracking of risk behaviours and factors through integration with devices; a wellness plan; access to a personal on-line health coach; goal-setting notifications; on-line community forums; and, circle of care access to information. The aim of this project is to evaluate the effects of VCRP (with integrated fitness tracker) compared to a standard, home-based CR program. The study will look at changes in: patient empowerment; health behaviours; risk factors; quality of life; clinical outcomes; and, costs. The study will improve our understanding of: patient and provider needs; program usability; and shared decision-making. Results will inform the use of e-health programs such as VCRP into healthcare settings to improve patient empowerment, shared decision-making, and the ability to integrate wearable monitors to improve health behaviours.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was hospitalized at the University of Ottawa Heart Institute (UOHI);
2. Patient has stable Coronary Heart Disease (CHD) or valvular disease;
3. Patient has been referred to Cardiac Rehabilitation (CR) and is a candidate an offsite program;
4. Patient has access to and regularly uses a smart phone, tablet or computer with Internet access;
5. Patient is ≥ 18 years of age (the age of consent in Ontario);
6. Patient is able to read and understand English or French (programs are available in both languages);
7. Patient is eligible for Ontario Health Insurance Plan (to permit linkage with administrative data housed at the Institute for Clinical Evaluative Sciences [ICES]);

Exclusion Criteria:

1. Patient was hospitalized for heart failure, congenital heart disease, transplant or arrhythmia within the last 6 months;
2. Patient, in the opinion of the medical advisor (Dr. Andrew Pipe), manifests illness that would preclude participation in the interventions (e.g. cognitive impairment, active drug or alcohol dependence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Patient Activation | Baseline - 22 weeks
  Patient activation will be measured by the Patient Activation Measure (PAM) questionnaire.This 10-item tool assesses the degree to which a patient is engaged or disengaged with their health and how likely they are to self-manage it.The total score of the tool classifies a participant into one of 4 categories; disengaged and overwhelmed (level 1), becoming aware but still struggling (level 2), taking action (level 3) and maintaining behaviors and pushing further (level 4). Higher levels mean participants are becoming better at, or have fully begun to self-manage their health behaviors.

SECONDARY OUTCOMES:
Tobacco smoking | Baseline - 22 weeks
  Participants will be asked 2 questions about tobacco smoking. The first asks about tobacco smoking in the last 6 months. The second asks about tobacco smoking in the last 7 days. If the participant has recently quit smoking we will ask for their quit date. This intervention is not providing smoking cessation counseling however, we are interested in participants cessation attempt as a health behavior change.
Physical activity | Baseline - 22 weeks
  Physical activity will be measured by pedometer. Participants will wear the pedometer for 7 days at baseline and again at 22 week follow up.
Dietary behaviors | Baseline - 22 weeks
  Dietary behaviors will be measured by the Starting the Conversation questionnaire. The questionnaire consists of 8 questions asking about frequency of fast food/snack consumption, fruit, vegetable, fat consumption, snacking and sodium intake. The participant's total score at baseline (sum of all answers, answers ranging from 0-2) will be compared to their total score at week 22. A change is considered a reduction in this score (0-16) between the two study time points. Higher values equate to a diet that could require a change in eating habits (reduction of salty foods or snacks, increase in vegetables/fruits).
Medication adherence | Baseline - 22 weeks
  Medication adherence will be assessed using the Medication Adherence Rating Scale (MARS). This is a 10 item questionnaire that generates a total score out of 10. The higher the score, the greater the adherence.
Blood pressure | Baseline - 22 weeks
  Blood pressure will be measured and recorded in millimeters of mercury. A high measured will be considered 140/90 or higher.
Low density lipoprotein cholesterol (LDL-C) | Baseline - 22 weeks
  LDL-C will be measured and reported in millimoles per litre (mmol/L). Measures < 3.5 mmol/L are considered desirable.
High density lipoprotein cholesterol (HDL-C) | Baseline - 22 weeks
  HDL-C will be measured and reported in millimoles per litre (mmol/L). Measures above 1.3 mmol/L are considered desirable.
Total cholesterol (TC) | Baseline - 22 weeks
  TC will be measured and reported in millimoles per litre (mmol/L). Measures less than 5.2 mmol/L are considered desirable.
Triglycerides | Baseline - 22 weeks
  Triglycerides will be measured and reported in millimoles per litre (mmol/L). Measures less than 5.2 mmol/L are considered desirable. Measures less than 1.7 mmol/L are considered desirable.
Glycated hemoglobin (A1C) | Baseline - 22 weeks
  Fasting A1C will be measured and reported in millimoles per litre (mmol/L). Measures between 4.0 to 7.0 mmol/L are considered desirable.
Waist circumference | Baseline - 22 weeks
  Waist circumference will be collected (measured in cm). A measurement of 88cm or more in women is considered high and is associated with health problems such as risk of developing type 2 diabetes, heart disease and high blood pressure.
Generic Quality of Life | Baseline - 22 weeks
  Generic health-related quality of life will be collected by the Short form Health Survey (SF-36, V1). This is a 36-item questionnaire assessing eight health concepts (physical functioning; role limitations because of physical health problems; bodily pain; social functioning; general mental health (psychological distress and psychological wellbeing); role limitations because of emotional problems; vitality (energy/fatigue); and general health perceptions). Questions are scored on a Likert scale which are then summed to a total between 0-100. Scores are then matched against norm tables.
  to produce raw scale scores for each health concept which are then transformed to a 0 - 100 scale
Health Related Quality of Life | Baseline - 22 weeks
  Disease specific quality of life will be measured using the Health-related quality of life questionnaire (HeartQoL). This is a 14 item questionnaire developed for use in patients with cardiac disease. There are 10 items related to physical health and 4 related to emotional health. Sub-scales are scored from 0 (poor quality of life) to 3 (better quality of life). Questions are summed to produce a total score.
Clinical outcomes - Re-hospitalization | Baseline - 52 weeks
  Re-hospitalization will be measured at 1-year. This will be accomplished by linking healh card numbers from study participants to administrative data housed at the Institute for Clinical Evaluative Sciences (ICES).
Clinical outcome - Health care utilization - Number of emergency room and physician visits | Baseline - 52 weeks
  The total number of emergency room visits and physician/specialist visits will be tallied at 1-year. This will be accomplished by linking health card numbers from study participants to administrative data housed at the Institute for Clinical Evaluative Sciences (ICES).
Clinical outcome - mortality | Baseline - 52 weeks
  Mortality will be measured at 1-year. This will be accomplished by linking healh card numbers from study participants to administrative data housed at the Institute for Clinical Evaluative Sciences (ICES).
Cost of Intervention | Fiscal year 2017 through study completion.
  The costs associated with delivering the VCRP and CMHP interventions will be collected during the study period. All costs will be expressed in Canadian dollars for the year 2017 and evaluated from the perspective of the healthcare system. Costs will be based on real resource use and will include the sum of the costs associated with assessments, coaching, and materials used (e.g., manuals, Garmin monitors).

OTHER OUTCOMES:
Patient Experiences with the VCRP Intervention and online Platform | Baseline - 22 weeks
  Patient's experiences will be assessed through focus group sessions. Participation is optional. Participants will be asked about their experiences with the VCRP, their acceptability and satisfaction with the VCRP, and suggestions for improvement. Participants will all be asked specific questions related to the VCRP platform but then given time to provide more general comments. The focus group questions will all be assembled by one of the Co-Investigators who has experience conducting focus group sessions. The Co-I will transcribe all focus group conversations and generate common themes. There are no score-able questionnaires being used during focus group sessions. These sessions are qualitative in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Mullen, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] CACPR 2020 Annual Meeting Abstracts. J Cardiopulm Rehabil Prev. 2020 Nov 1;40(6):E52-E57. doi: 10.1097/HCR.0000000000000561. No abstract available. PMID 33953036